CLINICAL TRIAL: NCT05185323
Title: Evaluation of the Effectiveness of Osteopathic Treatment on the Mother-newborn Dyad in the Event of Painful Breastfeeding in the Maternity Hospital Despite the Application of All Usual Aids: Randomized Interventional Study in Clusters in Two Parallel Arms Without Blinding. AMATOSTEO
Brief Title: Painful Breastfeeding and Osteopathic Treatment on the Mother-newborn Dyad
Acronym: AMATOSTEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2018/38
Record Dates: First submitted 2021-12-01; First posted 2022-01-11 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Painful Breastfeeding
Keywords: Osteopathic manipulative treatment; pain; breastfeeding
MeSH Terms: conditions — Pain; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding usual known aids and osteopathic treatment (Experimental): The osteopathic treatment consists of manual listening without intention, without thrust. The hands follow the spontaneous movements of the patients. The end of the treatment is perceived by an overall relief and a feeling of balance for the baby and his mother
  Interventions: Other: Breastfeeding usual known aids and osteopathic treatment
- Breastfeeding usual known aids (Active Comparator): Breastfeeding usual known aids in usual care
  Interventions: Other: Breastfeeding usual known aids

INTERVENTIONS:
Other: Breastfeeding usual known aids and osteopathic treatment — Breastfeeding usual known aids and osteopathic treatment
  Arms: Breastfeeding usual known aids and osteopathic treatment
Other: Breastfeeding usual known aids — Breastfeeding usual known aids
  Arms: Breastfeeding usual known aids

SUMMARY:
Pain during lactation is the first reason to stop breastfeeding. When usual known aids are ineffective, osteopathic treatment is a possible way to decrease the pain and improve the quality and the duration of lactation. The aim of this study is to compare usual known aids alone and usual known aids added to osteopathic treatment of the baby and the mother. The primary outcome is the lactation rate (exclusive or partial) at 1 month after birth

DETAILED DESCRIPTION:
Breastfeeding is recognized to be essential for childhood health and public health. The first reason to stop breastfeeding before the second month after birth is pain during lactation. The second reason to stop breastfeeding is back-to-work, generally two months after birth. Few years ago, osteopathic treatment has been introduced at maternity hospital of Bordeaux when usual known aids are ineffective. The osteopathic treatment is completely integrated in the maternity hospital of Bordeaux but no strong evaluation is available in literature. A pilot evaluation on 27 patients showed a good effectiveness of osteopathic treatment on breastfeeding at 1 months ½ after birth (85% of patients) Breast pain decreased or disappeared after the osteopathic treatment. Another evaluation showed a small rate of lactation (15% of patients) in a non treated group at 1 month ½. In the present study, osteopathic treatment will be added to usual known aids for 40 mother-newborn dyads when pain during lactation is greater than 7 (0 to 10 scale). The experimental group will be compared with 40 "non treated" mother-newborn dyads (only usual known aids in routine care). Among other, breastfeeding and pain during lactation will be evaluated at the maternity hospital discharge and will be repeated at 1 month after birth.

ELIGIBILITY:
Inclusion Criteria:

* Mother 18 yrs and older who chose to breast-feed (exclusive or not)
* Singleton newborn after 37 weeks of gestation, weighing at least 2500 g at birth, after 36 hours of life
* Pain during lactation greater than 7 (scale 0 to 10) in one or both breasts
* Usual known aids ineffective to reduce pain during lactation
* Mother speaking and understanding French
* Mother affiliated or beneficiary to a health system
* Signed informed consent.

Exclusion Criteria:

* Medical contraindication to osteopathic treatment (non stabilized infection, acute neurological pathology, tumor or cancer process, maternal psychiatric disorders)
* Severe congenitale malformation, especially not allowing normal lactation
* Patient under legal protection
* Persons deprived of their liberty by judicial or administrative decision

Min Age: 3 Days | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Proportion of women still breastfeeding | 1 month after birth
  Proportion of women still breastfeeding even if not exclusive

SECONDARY OUTCOMES:
Pain during lactation | 7 days, 1 month
  Pain at each breast during lactation after osteopathic treatment (analogic visual evaluation from 0-no pain to 10-extreme pain)
breastfeeding | 7 days, 1 month
  Proportion of women still breastfeeding even if not exclusive
Proportion of women still exclusive breastfeeding | 1 month
  Proportion of women still exclusive breastfeeding
Amount of artificial milk given per day | 1 month
  Amount of artificial milk given per day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elleau C, Missmahl C, Belcadi W, Aurillac-Lavignolle V, Sentilhes L. Evaluation of the effectiveness of osteopathic treatment on the mother-newborn dyad in the event of painful breastfeeding in a maternity hospital despite the application of all usual aids: randomized interventional trial in two parallel arms without blinding. Front Nutr. 2025 Apr 24;12:1577502. doi: 10.3389/fnut.2025.1577502. eCollection 2025. PMID 40342372